CLINICAL TRIAL: NCT01254513
Title: Randomized Phase II Study Evaluating the Feasibility of a Chemotherapy With Docetaxel-Prednisone in a Weekly Schedule or Every 3 Weeks, for Castration-resistant Metastatic Prostate Cancer Elderly Patients (>=75), "Vulnerable" or "Frail" , as Defined by the Criteria of the International Society of Geriatric Oncology (SIOG)
Brief Title: Feasibility of a Chemotherapy With Docetaxel-Prednisone for Castration-resistant Metastatic Prostate Cancer Elderly Patients
Acronym: GERICO10
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GERICO10/0910 (GetugP03)
Record Dates: First submitted 2010-10-26; First posted 2010-12-06 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Prostate Cancer
Keywords: Metastatic Prostate cancer; Elderly patients; Vulnerable and Frail (SIOG classification); castration-resistant
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Prednisone; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - Docetaxel every 3 weeks + Prednisone (Experimental): * Docetaxel: 60 mg/m²/day at C1 then 70 mg/m²/day for subsequent cycles every 3 weeks
  * Prednisone 10 mg/day continuously
  Interventions: Drug: Docetaxel every 3 weeks + Prednisone; Drug: Docetaxel weekly+ Prednisone
- Arm B - Docetaxel weekly + Prednisone (Experimental): * Docetaxel weekly 35 mg/m²/day on day 1 and day 8 of each cycle (J1 = J21)
  * Prednisone 10 mg/day continuously
  Interventions: Drug: Docetaxel weekly+ Prednisone

INTERVENTIONS:
Drug: Docetaxel every 3 weeks + Prednisone — * Docetaxel IV 60 mg/m²/d then IV 70 mg/m²/d for subsequent cycles every 3 weeks
  * Prednisone 10 mg/day continuously
  Other Names: TAXOTERE
  Arms: Arm A - Docetaxel every 3 weeks + Prednisone
Drug: Docetaxel weekly+ Prednisone — * Docetaxel weekly 35 mg/m²/day at day 1 and day 8 of each cycle (J1 = J21)
  * Prednisone 10 mg/day continuously
  Other Names: TAXOTERE

SUMMARY:
The objective of this study is to evaluate the feasibility of two different chemotherapy protocols with adjusted doses for patients aged 75 and over who often have medical problems other than prostate cancer. Patient will receive Docetaxel either every 3 weeks or weekly. In both cases, chemotherapy is combined with prednisone. The protocol will be considered feasible when patient will receive 6 cycles of chemotherapy (1 cycle = 3 weeks).

Additionally to this primary objective, efficacy will also be evaluated for both protocols as well as tolerance to treatment, quality of life and evolution of geriatric data.

DETAILED DESCRIPTION:
Standard management of castration-resistant metastatic prostate cancer is represented by chemotherapy with Docetaxel 75 mg/m² every 3 weeks combined with Prednisone since a symptomatic and overall survival benefit was demonstrated.

Although this benefit is independent of age in the study by Tannock (cut-off:69), it does not seem possible to extrapolate these results, obtained in a selected population, to the majority of patients we encounter in daily practice, >= 75 years old and / or unfit.

Retrospective studies have shown that chemotherapy was feasible, at standard or adapted doses in an unselected elderly population with good results in terms of tolerance and efficacy over symptoms.

Our study aims to evaluate prospectively the feasibility of a chemotherapy with Docetaxel/Prednisone administered every 3 weeks (60 mg / m² at D1C1 then 70 mg / m² at D1 for subsequent cycles if tolerance is good) or weekly (35mg / m² at D1 and D8 with Day 1 = Day 21) to patients >= 75 years old, evaluated by comprehensive geriatric assessment, belonging to group 2 "vulnerable" or to group 3 "frail" of the classification proposed by the International Society of Geriatric Oncology (SIOG).

Feasibility is defined as the possibility for a patient to receive 6 cycles of chemotherapy without withdrawal. Reasons for study withdrawal were defined by the GERICO Group and are the followings:

* stop or delay of chemotherapy > 2 weeks
* Necessity to reduce the dose of chemotherapy > 25 %
* febrile neutropenia or non-haematological grade 3 toxicity (except alopecia) according to NCI-CTCAE V4.0.
* Geriatric criterion (Activity of Daily Living (ADL) decrease >= 2 points)

The statistical methodology used is a double randomized phase II after stratification according to the SIOG criteria, based on a Simon Optimum plan.

A pharmacokinetic / pharmacodynamic study is associated to our project, based on a method of population pharmacokinetic. The aim is to highlight predictors of the haematological tolerance of this chemotherapy by evaluating clinical, geriatric and biological parameters.

The results of this study will support the terms of prescription of chemotherapy, in patients aged 75 and over, classified as "vulnerable" or "frail" regarding SIOG criteria, with defined geriatric assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 75
* Histologically proven prostate adenocarcinoma
* Metastatic disease, not pre-treated with chemotherapy refractory to castration
* Hormone refractory prostate cancer is defined as follows:

  * Patients with documented testosterone castration (<0.50 ng / ml)
  * Patient who received prior hormonal therapy (either orchidectomy or Luteinizing hormone-releasing hormone (LHRH) agonist alone or combined with an anti-androgen)
  * Patients should continue primary androgen suppression by LHRH agonist (in case of non-surgical castration)
  * For patients treated with anti-androgens prior to inclusion, a wash-out period is required (4 weeks for flutamide and nilutamide, 6 weeks for other products) as well as measured progression after anti-androgen discontinuation.
* Progressive disease under hormonotherapy, with progression defined by

Increase of PSA level (two consecutive increases of PSA compared to baseline with a minimum of one week between both measurements)

OR emergence of a new lesion

OR measurable progressive disease (increase of a previous measurable lesion >= 25% in cross section)

OR progressive bone metastases (defined only by the appearance of a new lesion on bone scan)

OR progressive symptoms (defined as cancer pain Grade 2 according to the NCI-CTC V4.0, despite level 2 analgesics intake).

* Patients of Groups 2 and 3 [ "vulnerable" and "frail"] of SIOG classification
* WHO Performance Status (PS) >= 3
* PSA >= 5 ng / ml
* Neutrophils >= 2.109 /L
* Platelets >= 100.109/L
* Haemoglobin ≥ 9 g/dl
* Bilirubin and SGOT / SGPT <1.5 x ULN (<= 2.5 x ULN if hepatic metastasis)
* creatinine <= 2.5 x ULN
* In case of previous palliative or analgesic radiotherapy, a minimum of 14 days must have elapsed between end of radiotherapy and inclusion into the study
* Previous treatment with bisphosphonates should be continued without change during the study treatment and can not be initiated either within 28 days prior to study entry or during the study
* Signed informed consent by patients, according to local regulations

Exclusion Criteria:

* "healthy" or "terminal illness" Groups according to the recommendations of International Society of Geriatric Oncology (SIOG)
* Concomitant or previous malignancy within 5 years prior the study (except basal or squamous in situ cell skin carcinoma)
* Presence of brain metastasis symptoms
* Prior treatment by intravenous radiopharmaceutical agent (e.g. Strontium 89, Samarium lexidronam) within 2 months before study entry
* Initiation of a bisphosphonate therapy within 28 days prior to randomisation
* Any concomitant anticancer treatment (radiotherapy, radiopharmaceutical agent, chemotherapy)
* Patients with uncontrolled infection
* Patients with peripheral neuropathy of grade> 1
* Patients medically unstable (e.g. unstable diabetes, uncontrolled hypertension or decompensated heart failure or myocardial infarct within 3 months)
* Gastro duodenal active ulcer
* Hypersensitivity to study drugs
* Treatment with any experimental drug within 30 days prior to or during the study
* Psychological, familial, sociological or geographical location conditions which do not allow medical monitoring and compliance with study protocol.
* Patients protected by the law or patients placed under protective supervision of adults

Min Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-12-09 (Actual); Primary Completion 2014-05-10 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Feasibility of 2 different protocols of Docetaxel chemotherapy | Up to 18 weeks (6 cycles of chemotherapy)
  Main criteria is the rate of patients receiving 6 cycles of treatment without experiencing any of the following criteria:
  * Stop or delay of chemotherapy > 2 weeks
  * Necessity to reduce the dose of chemotherapy > 25 %
  * Febrile neutropenia or non-haematological grade 3 toxicity (except alopecia)according to NCI-CTCAE V4.0
  * Geriatric criterion ( ADL decrease >= 2 points)

SECONDARY OUTCOMES:
Overall Survival | From randomization until death for any cause or last follow-up news (censored data)
  Overall Survival is defined as the time from randomization until death for any cause or last follow-up news (censored data).
Geriatric evaluation | At baseline, D1 of Cycle 1 and Cycle 4, at the end of treatment and at follow-up visits
  The impact of the chemotherapy will be evaluated on Comprehensive Geriatric Assessment :
  * Test de screening G8
  * Cumulative Illness Rating Scale(CIRSG)
  * Folstein Mini Mental State (MMS)
  * Activity of Daily Living (ADL)
  * Instrumental Activity of Daily Living (IADL)
  * Geriatric Depression Scale (GDS)
  * Mini Nutritionnal Assessment (MNA)
Number of patients with Adverse Events | At baseline, D1 of each cycle , at the end of treatment and at the follow-up visits
  Tolerance and safety will be assessed through recording of adverse events using NCI-CTCAE toxicity classification V4.0.
Quality of Life | At baseline, D1 of the Cycle 4, at the end of the treatment and at the follow-up visits
  The impact of the chemotherapy is evaluated on the European Organisation for Research and Treatment of Cancer (EORTC) Quality Of Life - Questionnaire - QLQ-C30
Vital signs measurement | At baseline, D1 of each cycle , at the end of treatment and at the follow-up visits
  Tolerance and safety will be assessed through vital signs measurement.
Prostate-specific antigen (PSA) measurements | At baseline, D1 of each cycle , at the end of treatment and at the follow-up visits
  Efficacy will be assessed through monitoring PSA values

CONTACTS AND LOCATIONS:
Overall Officials: Loic Mourey, Principal Investigator — Institut Claudius Regaud
Locations (31):
- France (31):
  - Clinique Claude Bernard, Albi
  - CHI Annemasse-Bonneville, Ambilly
  - Centre Paul Papin, Angers
  - CH de Blois, Blois
  - Institut Bergonie, Bordeaux
  - Centre Francois Baclesse, Caen
  - CH Intercommunal, Castres
  - Centre Hospitalier de Chambery, Chambéry
  - Centre Jean Perrin, Clermont-Ferrand
  - Clinique Sainte Marguerite, Hyères
  - Chd Vendee, La Roche-sur-Yon
  - Clinique Hartmann, Levallois-Perret
  - Centre Oscar Lambret, Lille
  - Hôpital Saint Vincent de Paul, Lille
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CHU Nimes, Nîmes
  - Chr Orleans, Orléans
  - Institut Curie/Claudius Regaud, Paris
  - Polyclinique Francheville, Périgueux
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier de La Region D'Annecy, Pringy
  - Institut Curie - Centre Rene Huguenin, Saint-Cloud
  - Ico - Centre Rene Gauducheau, Saint-Herblain
  - CH de Senlis, Senlis
  - Centre Paul Strauss, Strasbourg
  - Hôpitaux du Léman, Thonon-les-Bains
  - Institut Claudius Regaud, Toulouse
  - Polyclinique Du Parc, Toulouse
  - Clinique Saint Jean du Languedoc, Toulouse
  - Clinique Pasteur, Toulouse